CLINICAL TRIAL: NCT02580162
Title: Parents as Peer Interventionists in Treatment for Pediatric Weight Management
Brief Title: Success in Health: Impacting Families Together
Acronym: SHIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other); San Diego State University (Other)
Responsible Party: Principal Investigator, Brian Saelens, Professor of Pediatrics and Psychiatry and Behavioral Sciences, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK104863-01A1 (NIH)
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pro.Treatment, Not a Peer (Active Comparator): Families receive FBT for Pediatric Weight Management by Professionals interventionists and parents are NOT Peer Interventionists
  Interventions: Behavioral: FBT for Pediatric Weight Management by Professionals
- Pro.Treatment, Peer (Experimental): Families receive FBT for Pediatric Weight Management by Professionals and parents ARE Peer Interventionists
  Interventions: Behavioral: FBT for Pediatric Weight Management by Professionals; Behavioral: Peer Interventionists
- Peer Treatment, Not a Peer (Experimental): Families receive FBT for Pediatric Weight Management by Peers and parents are NOT Peer Interventionists
  Interventions: Behavioral: FBT for Pediatric Weight Management by Peers
- Peer Treatment, Peer (Experimental): Families receive FBT for Pediatric Weight Management by Peers and parents ARE Peer Interventionists
  Interventions: Behavioral: FBT for Pediatric Weight Management by Peers; Behavioral: Peer Interventionists

INTERVENTIONS:
Behavioral: FBT for Pediatric Weight Management by Professionals — This behavioral treatment includes behavioral skills training and accountability, including food and activity self-monitoring, goal setting, and home environment change. This 20 week treatment is adapted from our existing evidence-based interventions and is delivered by PROFESSIONAL interventionists.
  Arms: Pro.Treatment, Not a Peer; Pro.Treatment, Peer
Behavioral: FBT for Pediatric Weight Management by Peers — This behavioral treatment includes behavioral skills training and accountability, including food and activity self-monitoring, goal setting, and home environment change. This 20 week treatment is adapted from our existing evidence-based interventions and is provided by PEER interventionists.
  Arms: Peer Treatment, Not a Peer; Peer Treatment, Peer
Behavioral: Peer Interventionists — Parents who receive FBT complete 6 weeks of training and then serve as peer interventionists to a new group of families.
  Arms: Peer Treatment, Peer; Pro.Treatment, Peer

SUMMARY:
This study evaluates and compares the efficacy of professional versus peer-based delivery of family-based treatment for childhood overweight and obesity in elementary school aged children. Families will be randomized to receive treatment from professionals or to receive treatment from professionally-trained peer interventionists. Some parents will then be invited to serve as peer interventionists for the next group of families.

DETAILED DESCRIPTION:
The high prevalence of pediatric overweight and obesity in the U.S. necessitates the development of efficacious, but cost-effective and easily disseminable interventions that improve and sustain better pediatric weight outcomes. Accumulated evidence finds initial and long-term efficacy of moderate-to-high intensity (>25 contact hours) family-based treatment (FBT) for elementary school-aged children, but such treatment is prohibitively expensive because of high personnel costs (delivery by behavioral health professionals) and therefore limited in availability, reach, and impact. Very few overweight/obese children receive evidence-based treatment to improve their weight status or health.

The pilot data suggest a new model, peer-based delivery FBT with FBT-treated parents trained and subsequently delivering FBT to other families, is feasible and demonstrates initial efficacy. This delivery model could dramatically reduce FBT costs and increase FBT availability. Preliminary data also suggest that serving as a peer interventionist may also benefit the peers themselves and their children in better sustaining their own weight outcomes. The present study aims to provide a more definitive test of the short- and long-term efficacy of peer- versus professionally-delivered FBT on child weight outcomes. Embedded in this comparison is an examination of the feasibility of peer-based FBT delivery, investigating the impact of serving as a peer interventionist on the peers' own and their child's long- term weight status, and a more comprehensive examination of differential costs of professional- versus peer- based FBT delivery.

The present study will also test potential dissemination and sustainability by examining the efficacy of peer-delivered FBT among peer interventionists who themselves received FBT from other peers and not from professional interventionists. Moderation of treatment outcome is also examined, focusing on peer interventionist and child characteristics. This multi-phase trial will enroll 304 families with 7-11 year old overweight/obese children in multiple sites throughout the region, and include short-term (post-treatment) and long-term (up through 1 year after treatment cessation) assessments. This investigation of an innovative approach that could significantly reduce FBT delivery costs, while also improving the maintenance of treatment effects, is critical to improving the health of the many already overweight children at risk for chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Child age: 7-11 years at time of enrollment
* Overweight child: at or above 85th percentile for age- and gender-specific BMI.
* At least one overweight parent (BMI≥ 25.0).
* Parent is willing and able to actively participate in treatment including willingness to serve as a peer interventionist following treatment.
* Must live within 50 miles of the treatment center.

Exclusion Criteria:

* Current enrollment in another weight control program for the participating child or parent.
* The participating parent is pregnant.
* Thought disorder, suicidality, or substance abuse disorder in either the participating parent or the participating child.
* Inability of the child to comprehend English at a 1st-grade level or participating parent to comprehend English at an 8th-grade level.
* Physical disability or illness in either the participating parent or the child that precludes moderate intensity physical activity.
* Medication regimen for the child that affects his or her weight.
* Conditions known to promote obesity in the participating child (e.g. Prader-Willi).
* Diagnosed eating disorder (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder) in either parent (participating and nonparticipating) and/or the participating child.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Child BMI z-score | Baseline, 20 Weeks (post treatment), 6 and 12 months post treatment
  BMI will be calculated as kg/m2 and children's BMI z-scores will be calculated using CDC growth charts.

SECONDARY OUTCOMES:
Costs of Peer Versus Professional Treatment | 20 weeks
  Direct and indirect costs of associated with intervention using peer or professional interventionists. Direct costs will be estimated using hours spent providing treatment of both peers and professionals who will track their time using an online application. Costs associated with hours spent will be based on professional salaries or stipends provided to peer interventionists.
Change in Parent BMI | Baseline, 20 Weeks (post treatment), 6 and 12 months post treatment
  BMI of parent will be calculated as kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Saelens, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States